CLINICAL TRIAL: NCT06628700
Title: Burden Fatty Liver Among Acute Ischemic Cerebral Stroke Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mostafa Gamal Atef El-sayed, Resident doctor, Assiut University
Other Study IDs: Fatty liver
Record Dates: First submitted 2024-10-03; First posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Fatty Liver; Acute Ischemic Cerebral Stroke
Keywords: Fatty liver; Acute ischemic cerebral stroke; Hepatic steatosis
MeSH Terms: conditions — Fatty Liver

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 20 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
1. Assess frequency of hepatic steatosis among patients in patients with Ischemic stroke without previous risk factors
2. Assess outcomes morbidity and mortality ischemic stroke in correlation with hepatic steatosis .

DETAILED DESCRIPTION:
Fatty liver disease, encompassing both alcoholic and non-alcoholic variants, is a growing health concern worldwide, with prevalence rates soaring in parallel with obesity and diabetes epidemics. The estimated global incidence of NAFLD alone is 47 cases per 1,000 people, with a higher rate observed in males than females. Among adults worldwide, the estimated prevalence of NAFLD is 32%, with a higher prevalence in males (40%) compared to females (26%), making it the most common liver disorder. The hazards of fatty liver disease extend beyond the liver itself .The condition is characterized by the accumulation of excess fat in liver cells, which can progress to more severe liver diseases, such as steatohepatitis, fibrosis, cirrhosis, and hepatocellular carcinoma.

Early assessment and diagnosis of liver steatosis are crucial for managing and mitigating the risks associated with FLD. Non-invasive methods, such as elastography combined with the Controlled Attenuation Parameter (CAP) score, have emerged as effective tools for detecting and quantifying liver fat content. These methods offer a less invasive alternative to liver biopsies, providing reliable data to guide clinical decisions.

NAFLD is characterized by a proinflammatory and proatherogenic state that causes vascular inflammation and neurodegeneration, potentially leading to both clinical and subclinical cerebrovascular disease. Increasing epidemiological evidence links NAFLD to a higher risk and greater severity of stroke, independent of other vascular risk factors.Additionally, studies suggest NAFLD is involved in subclinical cerebrovascular diseases, such as carotid atherosclerosis which is characterized by the build-up of plaques in the carotid arteries. Patients with NAFLD exhibited greater carotid atherosclerosis .

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed ischemic cerebral stroke exceeding of window phase without obvious risk factors.
* patients above 18 years.
* patients below 60 years.

Exclusion Criteria:

* patients have obvious risk factors including: smoking, DM , Hypertension ,renal patients , cardiovascular diseases (AF , valvular disease ,reduced systolic function ,chronic HCV ,HBV).
* patients below 18 years.
* patients above 60 years.
* patients refused to contribute to this study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Newly diagnosed ischemic cerebral stroke patients exceeding of window phase without obvious risk factors.
Sampling Method: Non-Probability Sample
Enrollment: 97 (Estimated)
Dates: Start 2024-10-10 (Estimated); Primary Completion 2025-10-10 (Estimated); Study Completion 2025-11-10 (Estimated)

PRIMARY OUTCOMES:
Assess frequency of hepatic steatosis among patients in patients with Ischemic stroke without previous risk factors | Baseline

SECONDARY OUTCOMES:
Assess outcomes morbidity and mortality ischemic stroke in correlation with hepatic steatosis . | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Mostafa A Gamal, Principal Investigator — Assiut University; Noureldine A Abdelazeem, Study Director — Assiut University; Bahaa A Osman, Study Director — Assiut University

REFERENCES:
- [Background] Bonita R, Beaglehole R. Recovery of motor function after stroke. Stroke. 1988 Dec;19(12):1497-500. doi: 10.1161/01.str.19.12.1497. PMID 3201508
- [Background] DeGraba TJ, Hallenbeck JM, Pettigrew KD, Dutka AJ, Kelly BJ. Progression in acute stroke: value of the initial NIH stroke scale score on patient stratification in future trials. Stroke. 1999 Jun;30(6):1208-12. doi: 10.1161/01.str.30.6.1208. PMID 10356101
- [Background] Mughal MM, Khan MK, DeMarco JK, Majid A, Shamoun F, Abela GS. Symptomatic and asymptomatic carotid artery plaque. Expert Rev Cardiovasc Ther. 2011 Oct;9(10):1315-30. doi: 10.1586/erc.11.120. PMID 21985544
- [Background] Tahmasebpour HR, Buckley AR, Cooperberg PL, Fix CH. Sonographic examination of the carotid arteries. Radiographics. 2005 Nov-Dec;25(6):1561-75. doi: 10.1148/rg.256045013. PMID 16284135